CLINICAL TRIAL: NCT00000908
Title: Impact of Discontinuing PCP Prophylaxis in Subjects Receiving Antiretroviral Therapies Who Have Had Increases in CD4 Counts to > 200 Cells/mm3
Brief Title: A Study to Evaluate the Impact of Stopping Treatment for the Prevention of Pneumonia in HIV-Positive Patients Receiving Anti-HIV Drugs Who Have Increased CD4 Cell Counts
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: ACTG 888
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-02

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Pneumonia, Pneumocystis carinii; Antiviral Agents; CD4 Lymphocyte Count; RNA, Viral
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; AIDS-Related Opportunistic Infections

STUDY DESIGN:
Observational Model: Natural History

SUMMARY:
The purpose of this study is to see how often Pneumocystis carinii pneumonia (PCP) occurs in HIV-positive patients who have stopped taking medications that help prevent PCP.

The risk of developing PCP may be decreased when an HIV-positive patient's CD4 cell counts (cells of the immune system which fight infection) are more than 200 cells/mm3. This study looks at whether it is acceptable to stop PCP prevention treatment in these patients.

DETAILED DESCRIPTION:
The risk of developing PCP may be decreased with treatment-induced recovery of CD4 counts to > 200 cells/mm3. Few data exist to confirm or negate the continued necessity of PCP prophylaxis for such patients. This study will assess the effects of discontinuing therapy.

Subjects are asked to discontinue PCP prophylaxis if antiretroviral therapy has resulted in a sustained CD4 increase greater than 200 cells/mm3 on two measurements at least 12 weeks apart. They will be evaluated for symptoms and CD4 counts every 8 weeks as well as plasma for HIV-RNA every 16 weeks for 18 months. Subjects whose CD4 count falls to less than 150 cells/mm3 or between 150 and 200 cells/mm3 will have the CD4 count re-evaluated immediately or within 4 weeks. If the second CD4 count is less than 200 cells/mm3 for either case, conventional PCP prophylaxis will be resumed and the subject will be followed on study. Subjects will be followed during study by physical exams and laboratory tests at Weeks 4, 8, and every 8 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive.
* Have had 1 CD4 cell count of less than 100 cells/mm3 and have never had PCP, or have had at least 2 CD4 cell counts over 200 cells/mm3 and have had PCP within 6 months prior to study entry.
* Have received PCP prevention medication within 3 months of study entry.
* Are at least 13 years old (need consent if under 18).
* Are taking anti-HIV (antiretroviral) medication at study entry.

Exclusion Criteria

You will not be eligible for this study if you:

* Have active PCP or symptoms of PCP within 2 weeks of study entry.
* Have a fever lasting more than 2 weeks.
* Have oral candidiasis (thrush).

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250

CONTACTS AND LOCATIONS:
Overall Officials: Susan Koletar, Study Chair; Alison Heald, Study Chair; Robert Murphy, Study Chair
Locations (54):
- United States (53):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Kaiser Foundation Hosp, Harbor City, California
  - Kaiser Permanente LAMC, Los Angeles, California
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - Willow Clinic, Menlo Park, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - San Francisco AIDS Clinic / San Francisco Gen Hosp, San Francisco, California
  - San Francisco Gen Hosp, San Francisco, California
  - Santa Clara Valley Med Ctr / AIDS Community Rsch Consortium, San Jose, California
  - Marin County Specialty Clinic, San Rafael, California
  - San Mateo AIDS Program / Stanford Univ, Stanford, California
  - Stanford Univ Med Ctr, Stanford, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Howard Univ, Washington D.C., District of Columbia
  - Univ of Miami School of Medicine, Miami, Florida
  - Emory Univ, Atlanta, Georgia
  - Queens Med Ctr, Honolulu, Hawaii
  - Univ of Hawaii / Leahi Hosp, Honolulu, Hawaii
  - Northwestern Univ Med School, Chicago, Illinois
  - Cook County Hosp, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Louis A Weiss Memorial Hosp, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Division of Inf Diseases/ Indiana Univ Hosp, Indianapolis, Indiana
  - Methodist Hosp of Indiana / Life Care Clinic, Indianapolis, Indiana
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Boston Med Ctr, Boston, Massachusetts
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - Univ of Minnesota, Minneapolis, Minnesota
  - St Louis Regional Hosp / St Louis Regional Med Ctr, St Louis, Missouri
  - Univ of Nebraska Med Ctr, Omaha, Nebraska
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - Beth Israel Med Ctr, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Chelsea Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - St Mary's Hosp (Univ of Rochester/Infectious Diseases), Rochester, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Univ of Kentucky Lexington, Cincinnati, Ohio
  - Case Western Reserve Univ, Cleveland, Ohio
  - MetroHealth Med Ctr, Cleveland, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Philadelphia Veterans Administration Med Ctr, Philadelphia, Pennsylvania
  - Univ of Pennsylvania at Philadelphia, Philadelphia, Pennsylvania
  - Univ of Pittsburgh Med Ctr, Pittsburgh, Pennsylvania
  - Julio Arroyo, West Columbia, South Carolina
  - Univ of Washington, Seattle, Washington
- Univ of Puerto Rico, San Juan, Puerto Rico

REFERENCES:
- [Background] Koletar SL, Heald AE, Finkelstein D, Hafner R, Currier JS, McCutchan JA, Vallee M, Torriani FJ, Powderly WG, Fass RJ, Murphy RL; ACTG 888 Study Team. A prospective study of discontinuing primary and secondary Pneumocystis carinii pneumonia prophylaxis after CD4 cell count increase to > 200 x 106 /l. AIDS. 2001 Aug 17;15(12):1509-15. doi: 10.1097/00002030-200108170-00008. PMID 11504983